CLINICAL TRIAL: NCT01407094
Title: Establishing Moderators and Biosignatures of Antidepressant Response for Clinical Care (EMBARC) for Depression
Brief Title: Establishing Moderators and Biosignatures of Antidepressant Response for Clinical Care for Depression
Acronym: EMBARC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Madhukar H. Trivedi, Principal Investigator, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Other
Other Study IDs: STU 092010-151
Record Dates: First submitted 2011-07-25; First posted 2011-08-01 (Estimated); Results first posted 2018-12-26 (Actual); Last update posted 2018-12-26 (Actual); Status verified 2018-12

CONDITIONS: Depression
Keywords: Depression, Major Depressive Disorder, Mood Disorder
MeSH Terms: conditions — Depression; Depressive Disorder, Major; Mood Disorders | interventions — Sertraline

STUDY DESIGN:
Intervention Model Description: Patients were entered into Stage 1, treated with sertraline (Treatment A) or placebo (Treatment B), and used for the primary analysis which included the identification of potential mediators and moderators of response for these two treatments.
  In stage two, responders to Treatment A remained on sertraline, and non-responders were switched to bupropion (Treatment C). Responders to Treatment B remained on placebo, and non-responders were switched to sertraline (Treatment D).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Sertraline (Active Comparator): SSRI monotherapy
  Interventions: Drug: Sertraline
- Placebo (Placebo Comparator): Placebo control
  Interventions: Drug: Placebo
- Bupropion (Active Comparator): BupropionXL
  Interventions: Drug: BupropionXL

INTERVENTIONS:
Drug: Sertraline — 50-200mg/day
  Other Names: Zoloft
  Arms: Sertraline
Drug: Placebo — 1-4 pills per day
  Arms: Placebo
Drug: BupropionXL — 150-450 mg/day
  Other Names: WelbutrinXL
  Arms: Bupropion

SUMMARY:
This study will examine multiple carefully selected clinical and biological markers, using both existing state-of-the-art technologies as well as pioneering, innovative approaches. The study is designed to identify moderators and mediators of treatment response for depression in order to specify a biosignature of treatment response for depression. Evaluation of the usefulness of these markers in a carefully conducted clinical trial comparing an antidepressant to placebo will assist in developing a Depression Treatment Response Index (DTRI) to help clinicians match treatments to patients with MDD, resulting in timely selection of treatments best suited for individual patients and thus approaching personalized treatment. The resulting index provides a truly novel means of synthesizing the contribution of key clinical and biological parameters in an easy to use tool for clinical care.

DETAILED DESCRIPTION:
The current study is designed to identify biomarkers for the prediction of differential treatment outcomes between the SSRI antidepressant sertraline (SERT) and placebo (PBO) in a randomized trial for patients with MDD. In addition, a second stage will collect data to explore moderators and mediators of treatment outcomes between pharmacologically distinct active treatment arms: sertraline (SERT), a serotonergic antidepressant or bupropion (BUP), a nonserotonergic antidepressant. To reduce biologic heterogeneity, we will only enroll patients with early onset of DSM IV MDD (before age 30) because these criteria in probands have been shown to be associated with increased familial loading in families. Patients will also have recurrent MDD with 2 or more recurrences (including current episode). Additionally, patients will be required to have a current symptom severity score of 14 or more on the Quick Inventory of Depressive Symptomatology - Self Report (QIDS-SR), both at study screening and at the randomization (baseline) visit. In the first stage, patients will receive an 8-week course of treatment in one of the two study arms. As part of the Sequential Multiple Assignment Randomized Trial (SMART) design patients that have not achieved a response at the end of 8 weeks to their stage one treatment, defined by < 50% improvement on the Clinical Global Improvement scale (CGI), will be switched to Stage 2 treatment (8 weeks). Patients who have achieved satisfactory response (>= 50% improvement on the CGI) will be continued on treatment for an additional 8 weeks.

Specific Aims

Moderator Aims (Aim 1): To identify baseline clinical, neuroimaging, neurophysiological, and behavioral moderators of differential treatment outcome (mean symptom change and tolerability) for sertraline (SERT, a serotonergic antidepressant) versus placebo (PBO) for the treatment of MDD. Symptom change will be measured using the mean change from baseline in the 17-item Hamilton Rating Scale for Depression (HRSD17). Tolerability will be measured using the Frequency, Intensity, and Burden of Side Effects Rating (FIBSER) and the Treatment Emergent Symptom Scale (TESS).

Mediator Aims (Aim 2): To identify early phase (week 1) changes in neuroimaging, neurophysiological, and behavioral tasks as mediators of differential treatment outcomes (symptom change, tolerability) to SERT and PBO.

Main Treatment Effects Aim (Aim 3): To compare the 8-week outcomes of SERT vs. PBO using mixed model regression analysis to maximize power to discriminate treatment efficacy differences.

Primary Outcomes:

- 17-item Hamilton Rating Scale for Depression (HRSD17)

Secondary Outcomes:

- the Frequency, Intensity, and Burden Side Effects Rating (FIBSER)

ELIGIBILITY:
Inclusion Criteria:

* Adults, age 18-65
* Written informed consent obtained
* Outpatients with a current primary diagnosis of nonpsychotic recurrent or chronic MDD per the SCID-I
* QIDS-SR score of ≥ 14 at Screening Visit and Randomization (Baseline) Visit
* No failed antidepressant trials of adequate dose and duration, as defined by the MGH-ATRQ, in the current episode
* Agrees to, and is eligible for, all biomarkers procedures (EEG/psychological testing, MRI, and blood draws)

Exclusion Criteria:

* History of inadequate response (to trials at adequate dose for adequate duration) or poor tolerability to sertraline (SERT) or bupropion (BUP)
* Pregnant or breastfeeding
* Plan to become pregnant over the ensuing 12 months following study entry or are sexually active and not using adequate contraception
* History (lifetime) of psychotic depression, schizophrenia, bipolar (I, II, or NOS) disorder, schizoaffective disorder, or other Axis I psychotic disorder
* Current primary anxiety disorder diagnosis
* Meeting DSM-IV criteria for substance abuse in the last 2 months or substance dependence in the last 6 months (except for nicotine)
* Require immediate hospitalization for psychiatric disorder
* Have an unstable general medical condition (GMC) that will likely require hospitalization or to be deemed terminal (life expectancy < 6 months after study entry)
* Require medications for their GMCs that contraindicate any study medication
* Have epilepsy or other conditions requiring an anticonvulsant
* Receiving or have received during the index episode vagus nerve stimulation, ECT, or rTMS, or other somatic antidepressant treatments
* Currently taking any of the following exclusionary medications: antipsychotic medications, anticonvulsant medications, mood stabilizers, central nervous system stimulants, daily use of benzodiazepines or hypnotics, or antidepressant medication used for the treatment of depression or other purposes such as smoking cessation, since these agents may interfere with the testing of the major hypotheses under study. Nonexcluded concomitant medications are acceptable as long as their clinician determines that antidepressant treatment is safe and appropriate.
* Significant liver disease that would contraindicate any study medication
* Taking thyroid medication for hypothyroidism may be included only if they have been stable on the thyroid medication for 3 months
* Using agents that are potential augmenting agents (e.g., T3 in the absence of thyroid disease, SAMe, St. John's Wort, lithium, buspirone, Omega 3 fatty acids)
* Therapy that is depression specific, such as CBT or Interpersonal Psychotherapy of Depression (IPT) is not allowed during participation (participants can participate if they are receiving psychotherapy that is not targeting the symptoms of depression, such as supportive therapy, marital therapy).
* Subjects must be fluent in English and have the capacity to understand the nature of the study and sign the written informed consent since non-English speaking personnel are not available for this study, and the research instruments are not yet translated and validated in other languages.
* Currently actively suicidal or considered a high suicide risk
* Are currently enrolled in another study, and participation in that study contraindicates participation in the EMBARC study.
* Any reason not listed herein yet, determined by the site PI, medical personnel, or designee that constitutes good clinical practice and that would in the opinion of the site PI, medical personnel, or designee make participation in the study hazardous.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 296 (Actual)
Dates: Start 2011-07-29 (Actual); Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Madhukar H Trivedi, M.D., Principal Investigator — University of Texas Southwestern Medical Center; Patrick J McGrath, M.D., Principal Investigator — Columbia University; Myrna Weissman, Ph.D., Principal Investigator — Columbia University; Ramin Parsey, M.D., Principal Investigator — Columbia University; Maurizio Fava, M.D., Principal Investigator — Massachusetts General Hospital
Locations (4):
- United States (4):
  - Massachusetts General Hospital Boston, Boston, Massachusetts
  - University of Michigan Ann Arbor, Ann Arbor, Michigan
  - Columbia Univerisity New York City, New York, New York
  - UT Southwestern Medical Center Dallas, Dallas, Texas

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Chase HW, Fournier JC, Greenberg T, Almeida JR, Stiffler R, Zevallos CR, Aslam H, Cooper C, Deckersbach T, Weyandt S, Adams P, Toups M, Carmody T, Oquendo MA, Peltier S, Fava M, McGrath PJ, Weissman M, Parsey R, McInnis MG, Kurian B, Trivedi MH, Phillips ML. Accounting for Dynamic Fluctuations across Time when Examining fMRI Test-Retest Reliability: Analysis of a Reward Paradigm in the EMBARC Study. PLoS One. 2015 May 11;10(5):e0126326. doi: 10.1371/journal.pone.0126326. eCollection 2015. PMID 25961712
- [Background] Fournier JC, Chase HW, Greenberg T, Etkin A, Almeida JR, Stiffler R, Deckersbach T, Weyandt S, Cooper C, Toups M, Carmody T, Kurian B, Peltier S, Adams P, McInnis MG, Oquendo MA, McGrath PJ, Fava M, Weissman M, Parsey R, Trivedi MH, Phillips ML. Neuroticism and Individual Differences in Neural Function in Unmedicated Major Depression: Findings from the EMBARC Study. Biol Psychiatry Cogn Neurosci Neuroimaging. 2017 Mar;2(2):138-148. doi: 10.1016/j.bpsc.2016.11.008. Epub 2016 Dec 6. PMID 28983519
- [Background] Greenberg T, Chase HW, Almeida JR, Stiffler R, Zevallos CR, Aslam HA, Deckersbach T, Weyandt S, Cooper C, Toups M, Carmody T, Kurian B, Peltier S, Adams P, McInnis MG, Oquendo MA, McGrath PJ, Fava M, Weissman M, Parsey R, Trivedi MH, Phillips ML. Moderation of the Relationship Between Reward Expectancy and Prediction Error-Related Ventral Striatal Reactivity by Anhedonia in Unmedicated Major Depressive Disorder: Findings From the EMBARC Study. Am J Psychiatry. 2015 Sep 1;172(9):881-91. doi: 10.1176/appi.ajp.2015.14050594. Epub 2015 Jul 17. PMID 26183698
- [Background] Petkova E, Ogden RT, Tarpey T, Ciarleglio A, Jiang B, Su Z, Carmody T, Adams P, Kraemer HC, Grannemann BD, Oquendo MA, Parsey R, Weissman M, McGrath PJ, Fava M, Trivedi MH. Statistical Analysis Plan for Stage 1 EMBARC (Establishing Moderators and Biosignatures of Antidepressant Response for Clinical Care) Study. Contemp Clin Trials Commun. 2017 Jun;6:22-30. doi: 10.1016/j.conctc.2017.02.007. Epub 2017 Feb 24. PMID 28670629
- [Background] Pizzagalli DA, Webb CA, Dillon DG, Tenke CE, Kayser J, Goer F, Fava M, McGrath P, Weissman M, Parsey R, Adams P, Trombello J, Cooper C, Deldin P, Oquendo MA, McInnis MG, Carmody T, Bruder G, Trivedi MH. Pretreatment Rostral Anterior Cingulate Cortex Theta Activity in Relation to Symptom Improvement in Depression: A Randomized Clinical Trial. JAMA Psychiatry. 2018 Jun 1;75(6):547-554. doi: 10.1001/jamapsychiatry.2018.0252. PMID 29641834
- [Background] Trivedi MH, South C, Jha MK, Rush AJ, Cao J, Kurian B, Phillips M, Pizzagalli DA, Trombello JM, Oquendo MA, Cooper C, Dillon DG, Webb C, Grannemann BD, Bruder G, McGrath PJ, Parsey R, Weissman M, Fava M. A Novel Strategy to Identify Placebo Responders: Prediction Index of Clinical and Biological Markers in the EMBARC Trial. Psychother Psychosom. 2018;87(5):285-295. doi: 10.1159/000491093. Epub 2018 Aug 15. PMID 30110685
- [Background] Trivedi MH, McGrath PJ, Fava M, Parsey RV, Kurian BT, Phillips ML, Oquendo MA, Bruder G, Pizzagalli D, Toups M, Cooper C, Adams P, Weyandt S, Morris DW, Grannemann BD, Ogden RT, Buckner R, McInnis M, Kraemer HC, Petkova E, Carmody TJ, Weissman MM. Establishing moderators and biosignatures of antidepressant response in clinical care (EMBARC): Rationale and design. J Psychiatr Res. 2016 Jul;78:11-23. doi: 10.1016/j.jpsychires.2016.03.001. Epub 2016 Mar 15. PMID 27038550
- [Background] Trombello JM, Pizzagalli DA, Weissman MM, Grannemann BD, Cooper CM, Greer TL, Malchow AL, Jha MK, Carmody TJ, Kurian BT, Webb CA, Dillon DG, McGrath PJ, Bruder G, Fava M, Parsey RV, McInnis MG, Adams P, Trivedi MH. Characterizing anxiety subtypes and the relationship to behavioral phenotyping in major depression: Results from the EMBARC study. J Psychiatr Res. 2018 Jul;102:207-215. doi: 10.1016/j.jpsychires.2018.04.003. Epub 2018 Apr 6. PMID 29689518
- [Background] Ulke C, Tenke CE, Kayser J, Sander C, Bottger D, Wong LYX, Alvarenga JE, Fava M, McGrath PJ, Deldin PJ, Mcinnis MG, Trivedi MH, Weissman MM, Pizzagalli DA, Hegerl U, Bruder GE. Resting EEG Measures of Brain Arousal in a Multisite Study of Major Depression. Clin EEG Neurosci. 2019 Jan;50(1):3-12. doi: 10.1177/1550059418795578. Epub 2018 Sep 5. PMID 30182751
- [Background] Webb CA, Trivedi MH, Cohen ZD, Dillon DG, Fournier JC, Goer F, Fava M, McGrath PJ, Weissman M, Parsey R, Adams P, Trombello JM, Cooper C, Deldin P, Oquendo MA, McInnis MG, Huys Q, Bruder G, Kurian BT, Jha M, DeRubeis RJ, Pizzagalli DA. Personalized prediction of antidepressant v. placebo response: evidence from the EMBARC study. Psychol Med. 2019 May;49(7):1118-1127. doi: 10.1017/S0033291718001708. Epub 2018 Jul 2. PMID 29962359
- [Derived] Chin Fatt CR, Minhajuddin A, Jha MK, Mayes T, Rush AJ, Trivedi MH. Data driven clusters derived from resting state functional connectivity: Findings from the EMBARC study. J Psychiatr Res. 2023 Feb;158:150-156. doi: 10.1016/j.jpsychires.2022.12.002. Epub 2022 Dec 27. PMID 36586213
- [Derived] Jha MK, Schatzberg A, Minhajuddin A, Chin Fatt C, Mayes TL, Trivedi MH. Cross-Sectional Associations Among Symptoms of Pain, Irritability, and Depression and How These Symptoms Relate to Social Functioning and Quality of Life: Findings From the EMBARC and STRIDE Studies and the VitalSign6 Project. J Clin Psychiatry. 2021 Apr 13;82(3):20m13740. doi: 10.4088/JCP.20m13740. PMID 34000130
- [Derived] Jha MK, Fava M, Minhajuddin A, Chin Fatt C, Mischoulon D, Cusin C, Trivedi MH. Association of anger attacks with suicidal ideation in adults with major depressive disorder: Findings from the EMBARC study. Depress Anxiety. 2021 Jan;38(1):57-66. doi: 10.1002/da.23095. Epub 2020 Oct 10. PMID 33038902
- [Derived] Chin Fatt CR, Cooper C, Jha MK, Aslan S, Grannemann B, Kurian B, Greer TL, Fava M, Weissman M, McGrath PJ, Parsey RV, Etkin A, Phillips ML, Trivedi MH. Dorsolateral Prefrontal Cortex and Subcallosal Cingulate Connectivity Show Preferential Antidepressant Response in Major Depressive Disorder. Biol Psychiatry Cogn Neurosci Neuroimaging. 2021 Jan;6(1):20-28. doi: 10.1016/j.bpsc.2020.06.019. Epub 2020 Jul 8. PMID 32921587
- [Derived] Jha MK, Minhajuddin A, Chin Fatt C, Trivedi MH. Improvements in irritability with sertraline versus placebo: Findings from the EMBARC study. J Affect Disord. 2020 Oct 1;275:44-47. doi: 10.1016/j.jad.2020.06.021. Epub 2020 Jun 26. PMID 32658822
- [Derived] Rolle CE, Fonzo GA, Wu W, Toll R, Jha MK, Cooper C, Chin-Fatt C, Pizzagalli DA, Trombello JM, Deckersbach T, Fava M, Weissman MM, Trivedi MH, Etkin A. Cortical Connectivity Moderators of Antidepressant vs Placebo Treatment Response in Major Depressive Disorder: Secondary Analysis of a Randomized Clinical Trial. JAMA Psychiatry. 2020 Apr 1;77(4):397-408. doi: 10.1001/jamapsychiatry.2019.3867. PMID 31895437
- [Derived] Chin Fatt CR, Jha MK, Cooper CM, Fonzo G, South C, Grannemann B, Carmody T, Greer TL, Kurian B, Fava M, McGrath PJ, Adams P, McInnis M, Parsey RV, Weissman M, Phillips ML, Etkin A, Trivedi MH. Effect of Intrinsic Patterns of Functional Brain Connectivity in Moderating Antidepressant Treatment Response in Major Depression. Am J Psychiatry. 2020 Feb 1;177(2):143-154. doi: 10.1176/appi.ajp.2019.18070870. Epub 2019 Sep 20. PMID 31537090
- [Derived] Cooper CM, Chin Fatt CR, Jha M, Fonzo GA, Grannemann BD, Carmody T, Ali A, Aslan S, Almeida JRC, Deckersbach T, Fava M, Kurian BT, McGrath PJ, McInnis M, Parsey RV, Weissman M, Phillips ML, Lu H, Etkin A, Trivedi MH. Cerebral Blood Perfusion Predicts Response to Sertraline versus Placebo for Major Depressive Disorder in the EMBARC Trial. EClinicalMedicine. 2019 May 18;10:32-41. doi: 10.1016/j.eclinm.2019.04.007. eCollection 2019 Apr. PMID 31193824
- [Derived] Pillai RLI, Huang C, LaBella A, Zhang M, Yang J, Trivedi M, Weissman M, McGrath P, Fava M, Kurian B, Cooper C, McInnis M, Oquendo MA, Pizzagalli DA, Parsey RV, DeLorenzo C. Examining raphe-amygdala structural connectivity as a biological predictor of SSRI response. J Affect Disord. 2019 Sep 1;256:8-16. doi: 10.1016/j.jad.2019.05.055. Epub 2019 May 28. PMID 31158720
- [Derived] Whitton AE, Webb CA, Dillon DG, Kayser J, Rutherford A, Goer F, Fava M, McGrath P, Weissman M, Parsey R, Adams P, Trombello JM, Cooper C, Deldin P, Oquendo MA, McInnis MG, Carmody T, Bruder G, Trivedi MH, Pizzagalli DA. Pretreatment Rostral Anterior Cingulate Cortex Connectivity With Salience Network Predicts Depression Recovery: Findings From the EMBARC Randomized Clinical Trial. Biol Psychiatry. 2019 May 15;85(10):872-880. doi: 10.1016/j.biopsych.2018.12.007. Epub 2018 Dec 19. PMID 30718038
- [Derived] Liao A, Walker R, Carmody TJ, Cooper C, Shaw MA, Grannemann BD, Adams P, Bruder GE, McInnis MG, Webb CA, Dillon DG, Pizzagalli DA, Phillips ML, Kurian BT, Fava M, Parsey RV, McGrath PJ, Weissman MM, Trivedi MH. Anxiety and anhedonia in depression: Associations with neuroticism and cognitive control. J Affect Disord. 2019 Feb 15;245:1070-1078. doi: 10.1016/j.jad.2018.11.072. Epub 2018 Nov 14. PMID 30699849

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Final enrollment Stage 1: 296 (146 SERT, 150 PBO). Individuals who responded to their Stage 1 treatment remained on that treatment in Stage 2. Individuals who did not respond to their Stage 1 treatment were switched to a different treatment in Stage 2.
Groups:
- BupropionXL: BupropionXL
  150-450 mg/day
  Other names: WelbutrinXL
Period: Stage 1
Arm/Group | Sertraline | Placebo | BupropionXL
Started | 146 (Stage 1 Sertraline (SERT): 34 exited) | 150 (Stage 1 Placebo (PBO): 27 exited.) | 0 (Bupropion (BUP) was used only in Stage 2 for non-responders to SERT.)
Completed | 112 (One participant completed Stage 1 but did not continue to Stage 2.) | 123 (Four participants completed Stage 1 but did not continue to Stage 2.) | 0
Not Completed | 34 | 27 | 0
Period: Stage 2
Arm/Group | Sertraline | Placebo | BupropionXL
Started | 134 (Stage 2 SERT includes Stage 1 SERT responders (n=61) and Stage 1 PBO non-responders (n=73).) | 46 (Stage 2 PBO includes Stage 1 PBO responders (n=47); 1 early exit (n=46).) | 53 (Stage 2 BUP includes Stage 1 SERT non-responders (n=54); 1 early exit (n=53).)
Completed | 113 | 35 | 38
Not Completed | 21 | 11 | 15

BASELINE CHARACTERISTICS:
Population: Stage 1 is made up of Treatment A (SERT) and Treatment B (PBO). Non-responders to Treatment A were switched in Stage 2 to BUP, and non-responders in Treatment B were switched to SERT. Between randomization and baseline, 3 participants didn't meet inclusion criteria, hence the discrepancy between official enrollment and baseline population numbers.
Groups:
- BupropionXL: BupropionXL
  150-450mg/day
- Total: Total of all reporting groups
Arm/Group | Sertraline | Placebo | BupropionXL | Total
Number analyzed (Participants) | 146 | 150 | 0 | 296
Age, Categorical [Count of Participants; unit: Participants] — Population: Of the 299 participants who were randomized, 3 were randomized but did not meet criteria, resulting in 296 who were randomized and assessed.
  Participants
    <=18 years | 6 | 4 |  | 10
    Between 18 and 65 years | 139 | 145 |  | 284
    >=65 years | 1 | 1 |  | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.2 (13.8) | 36.9 (12.8) |  | 37.05 (13.3)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Measure Analysis Population Description: Of the 299 participants who were randomized, 3 were randomized but did not meet criteria, resulting in 296 who were randomized and assessed
  Participants
    Female | 102 | 92 |  | 194
    Male | 44 | 58 |  | 102
Region of Enrollment [Number; unit: participants]
  United States | 146 | 150 |  | 296

OUTCOME MEASURES:

1. Primary Outcome: Hamilton Rating Scale for Depression
Description: The Hamilton Rating Scale for depression is a measure of depressive severity (HAM-D17; HDRS)
  * Scores range from 0-52
  * Lower scores indicate less depressive symptomatology, and so are the more desirable.
Time Frame: Week 8
Population: Note subjects in the efficacy trial were those that completed 8 weeks of treatment, 115 in the sertraline group, and 123 in the placebo group. SERT had 34 wash-outs, PBO had 27.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sertraline | Placebo | BupropionXL
Number analyzed (Participants) | 146 | 150 | 0
units on a scale | 11.06 (6.71) | 12.52 (7.68) |

ADVERSE EVENTS:
Time Frame: 8 weeks for each Stage (1 and 2)
Description: For both Serious and Other adverse events: SERT total is the sum of Stages 1 or 2, Treatment A plus Treatment D (210+73); PBO total is the sum of Stages 1 or 2, Treatment B (150+46). BUP was only used during Stage 2 (Treatment C).
Groups:
- BupropionXL: BupropionXL
  150-450 mg/day
Arm/Group | Sertraline | Placebo | BupropionXL
Serious Adverse Events (participants affected / at risk) | 10/283 | 7/196 | 1/53
Other Adverse Events (participants affected / at risk) | 233/283 | 89/196 | 27/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sertraline (N=283) | Placebo (N=196) | BupropionXL (N=53)
ER Visit (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) — Type-I Diabetes with brittle blood sugar control; hospital admin w/ ketoacidosis
ER Visit (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) — ER visit with diagnosis of acute cholecystitis
ER Visit (General disorders) | 1 (1) | 0 (0) | 0 (0) — ER visit with fever
Suicidality (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) — Emergent suicidality
ER Visit (General disorders) | 1 (1) | 0 (0) | 0 (0) — Chest pain with emergency hospitalization; diagnosis of non-cardiac chest pain
Suicidality (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) — Involuntary hospitalization for suicidality
Suicidality (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) — Worsening depression, suicidal ideation
Panic attack (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) — Panic attack, arrested
Panic attack (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) — Panic attack
Pregnancy (Reproductive system and breast disorders) | 0 (0) | 2 (2) | 0 (0) — Became pregnant
ER Visit (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) — Chest pain with emergency hospitalization
ER Visit (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) — Worsening depression, suicidal ideation to ER
Suicidality (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) — Hospitalization for suicidality
Pregnancy (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) — Exited study due to pregnancy on 9/16/12 and gave birth to microcephalic child on 5/7/13
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) — Seizure
Hospitalization (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) — Worsening depression, suicidal ideation; psych hospitalization
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sertraline (N=283) | Placebo (N=196) | BupropionXL (N=53)
Diarrhea (Gastrointestinal disorders) | 34 (34) | 11 (11) | 2 (2)
Dizziness (General disorders) | 12 (12) | 6 (6) | 6 (6)
Fatigue (General disorders) | 13 (13) | 2 (2) | 1 (1)
Dry Mouth (General disorders) | 33 (33) | 8 (8) | 0 (0)
Headaches (General disorders) | 41 (41) | 46 (46) | 9 (9)
Insomnia (General disorders) | 30 (30) | 3 (3) | 1 (1)
Nausea (General disorders) | 57 (57) | 10 (10) | 5 (5)
Palpitations (Cardiac disorders) | 13 (13) | 3 (3) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No